CLINICAL TRIAL: NCT01915108
Title: Optimal Effect-site Concentration of Remifentanil for Inhibiting Response to Laryngeal Mask Airway (LMA) Removal During Emergence From Sevoflurane-remifentanil Anesthesia
Brief Title: Optimal Effect-site Concentration of Remifentanil for Inhibiting Response to Laryngeal Mask Airway (LMA) Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangjin Park (Other)
Responsible Party: Sponsor-Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Organization: Yeungnam University College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: apsj1
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Respiratory Complication
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- group R0 (No Intervention): remifentanil Ce of 0 ng/ml
- group R0.5 (Active Comparator): remifentanil Ce of 0.5 ng/ml
  Interventions: Drug: Remifentanil
- group R1.0 (Active Comparator): remifentanil Ce of 1.0 ng/ml
  Interventions: Drug: Remifentanil
- group R1.5 (Active Comparator): remifentanil Ce of 1.5 ng/ml
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — All patients received a predetermined Ce of remifentanil by TCI according to their group assignments 10 minutes before the end of surgery (R0, remifentanil Ce of 0 ng/ml; R0.5, remifentanil Ce of 0.5 ng/ml; R1.0, remifentanil Ce of 1.0 ng/ml; R1.5, remifentanil Ce of 1.5 ng/ml).
  Other Names: remifentanil (ultiva)
  Arms: group R0.5; group R1.0; group R1.5

SUMMARY:
This study was designed to determine the optimal dose of remifentanil that can prevent the complications associated with the removal of LMA without delaying emergence.

DETAILED DESCRIPTION:
Patients were randomly assigned to one of four groups. All patients received a predetermined effect-site concentrations (Ce) of remifentanil by target-controlled infusion (TCI) according to their group assignments (R0, remifentanil Ce of 0 ng/ml; R0.5, remifentanil Ce of 0.5 ng/ml; R1.0, remifentanil Ce of 1.0 ng/ml; R1.5, remifentanil Ce of 1.5 ng/ml) from 10 minutes before the end of surgery to LMA removal. Airway complications (airway obstruction, desaturation, breath holding, and coughing), nausea, and vomiting were assessed during the emergence phase.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 or 2
* undergoing lower extremity surgery under general anesthesia

Exclusion Criteria:

* suspected difficult airways
* respiratory disease (chronic obstructive pulmonary disease, upper respiratory infection)
* body mass index > 30 kg/m2
* allergies to the study drugs
* a history of gastric reflux

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sangjin park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group R0 | Group R0.5 | Group R1.0 | Group R1.5
Started | 32 | 32 | 32 | 32
Completed | 30 (two patients were excluded from the study) | 29 (three patients were excluded from the study) | 31 (one patients were excluded from the study) | 30 (two patients were excluded from the study)
Not Completed | 2 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group R0 | Group R0.5 | Group R1.0 | Group R1.5 | Total
Number analyzed (Participants) | 30 | 29 | 31 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 31 | 30 | 120
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 16 | 15 | 62
  Male | 16 | 12 | 15 | 15 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events Following LMA Removal
Description: All patients received a predetermined Ce of remifentanil by TCI according to their group assignments from 10 minutes before the end of surgery to LMA removal. Adverse events such as coughing, airway obstruction, breath-holding, desaturation, nausea and vomiting were evaluated from the end of surgery until arrival in the post-anesthetic care unit.
Time Frame: from the end of surgery until arrival in the post-anesthetic care unit, an expected average of 15 minutes.
Measure: Number; unit: participants
Arm/Group | Group R0 | Group R0.5 | Group R1.0 | Group R1.5
Number analyzed (Participants) | 30 | 29 | 31 | 30
participants | 10 | 5 | 1 | 0

ADVERSE EVENTS:
Groups:
- Group R0: remifentanil Ce of 0 ng/ml
  Remifentanil: All patients received a predetermined Ce of remifentanil by TCI according to their group assignments 10 minutes before the end of surgery (R0, remifentanil Ce of 0 ng/ml; R0.5, remifentanil Ce of 0.5 ng/ml; R1.0, remifentanil Ce of 1.0 ng/ml; R1.5, remifentanil Ce of 1.5 ng/ml).
Arm/Group | Group R0 | Group R1.5 | Group R0.5 | Group R1.0
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30 | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 13/30 | 6/30 | 14/29 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group R0 (N=30) | Group R1.5 (N=30) | Group R0.5 (N=29) | Group R1.0 (N=31)
airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group R0 (N=30) | Group R1.5 (N=30) | Group R0.5 (N=29) | Group R1.0 (N=31)
breath holding (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 6 (6) | 14 (14) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes